CLINICAL TRIAL: NCT05652088
Title: The Role of the Gastrointestinal-associated Lymphoid Tissue in the Cure of HIV Infection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Francesca Cossarini, Assistant Professor of Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY-22-01294
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Colonoscopy

STUDY DESIGN:
Intervention Model Description: All subjects receiving therapies with the potential for HIV cure who agree to participate in this study, will undergo a colonoscopy to obtain tissue samples for research assays before and after receiving such treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with HIV Therapy (Experimental): Subjects receiving therapies with the potential for HIV cure
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy — Colonoscopy is a procedure where an instrument called colonoscope is inserted through the rectum to look at the entire internal surface of the intestine. Participants will be placed on a stretcher on the left side. A colonoscope will be advanced into the colon and into the terminal ileum. The entire procedure should take approximately 40 minutes

SUMMARY:
The objective of this study is to understand the effects of HIV cure strategies on the virus and immune cells that reside within the gastrointestinal tract. Subjects receiving therapies with the potential for HIV cure will undergo a colonoscopy to obtain gastrointestinal tissue for research assays. This study will test whether receiving these therapies will induce changes in the immune cells in the gastrointestinal tract and reduce the tissue-associated HIV viral levels.

DETAILED DESCRIPTION:
After almost forty years from its first discovery, Human Immunodeficiency Virus (HIV) infection remains uncurable. The major obstacle to a cure for HIV infection is the integration of HIV into the host genome and its persistence in populations of long-lived immune cells subsets. These long-lived resting cells represent a reservoir of transcriptionally silent HIV and they are mostly localized in the secondary lymphoid tissue and the gastrointestinal associated lymphoid tissue (GALT).

The most promising HIV cure strategies relay on molecules which can induce enhanced immune responses through antibody mediated effects such as antibody-dependent cellular cytotoxicity (ADCC) and phagocytosis (ADCP) as well as enhanced CD8+ T cells activity.

The specific purpose of this study is to evaluate whether the proposed treatment strategies for HIV cure, can induce changes in the gastrointestinal associated immune system (GALT) effector immune cells such as NK cells, cytotoxic CD8+ T Cells and whether treatment with these molecules leads to changes in the amount of tissue-associated HIV virus within the GALT. The results from the proposed study will inform on the ability of these molecules to exert their effect on this critical site of HIV latency and persistence and thus advance the field on their HIV cure potential.

Subjects receiving treatment with the potential for HIV cure will undergo a colonoscopy to obtain gastrointestinal tissue for research assays. The research proposal will test the hypothesis of whether these molecules are able to induce changes in the immune cells in the gastrointestinal tract and reduce the tissue-associated HIV viral levels.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and lifestyle considerations and availability for the duration of the study
* Males and females; Age 18-75
* Chronic HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load
* Receiving treatment with a molecule with the potential for HIV cure
* Willingness and ability to undergo colonoscopy twice during the study timeframe

Exclusion Criteria:

* Known coagulopathy or altered coagulation studies
* Concomitant pregnancy of plans for pregnancy during the study period
* Concomitant Inflammatory Bowel Disease, Diarrheal disease or other gastrointestinal disease that might alter the intestinal mucosal tissue
* Concomitant sexually transmitted infection
* Any other condition which in the opinion of investigators would impede competence, compliance or possibly hinder completion of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in HIV tissue viral load | End of the study (at month one) compared to baseline
  Change in HIV in tissue-associated HIV RNA viral load at the end of the study at month one compared to baseline

SECONDARY OUTCOMES:
Change in number of Cytotoxic T cells | End of the study (at month one) compared to baseline
  Change in number of tissue-associated cytotoxic T cells at the end of the study (at month one) period compared to baseline
Change in number of NK Cells | End of the study (at month one) compared to baseline
  Change in number of tissue-associated NK cells at the end of the study (at month one) period compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Cossarini, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD at this time.